CLINICAL TRIAL: NCT00360906
Title: Omega-3 Fatty Acid Treatment in Multiple Sclerosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: The Multiple Sclerosis National Competence Centre (Unknown); The Norwegian Multiple sclerosis Society (Unknown); Pronova BioPharma (Industry); Serono Nordic (Unknown); Amersham Health (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NSD-10842; OFAMS, REK VEST, 005.04
Record Dates: First submitted 2006-08-04; First posted 2006-08-07 (Estimated); Last update posted 2006-08-07 (Estimated); Status verified 2006-08

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: RRMS; Omega-3; Treatment
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Fatty Acids, Omega-3

INTERVENTIONS:
Drug: Triomar™ (omega-3 fatty acids)

SUMMARY:
Based on previous clinical studies indicating beneficial treatment effects of omega-3 fatty acids in multiple sclerosis, and the increasing evidence of anti-inflammatory effects of omega-3 fatty acids, this study aims to evaluate treatment effects of concentrated omega-3 fatty acids (Triomar™) in MS, both as monotherapy and in combination with standard immunomodulatory therapy defined as interferon-beta 1a (Rebif™).

DETAILED DESCRIPTION:
Patients with relapsing-remitting multiple sclerosis with evidence of disease activity defined as at least one relapse or at least one new MRI lesion during the year prior to inclusion will be included in the study.

Eligible patients will be randomised for daily treatment with either oral omega-3 fatty acid (Triomar™) or placebo. After six months all patients will in addition receive interferon-beta 1a (Rebif™) 44 mcg subcutaneous three times per week for another 18 months.

The patients will undergo monthly contrast enhanced MRI for the first nine months and thereafter at months 12 and 24. They will also be examined by clinical and laboratory tests at six months intervals in addition to month 9 (3 months after start of IFNB treatment). Fatigue and QoL registration will be performed at baseline and at months 6, 12 and 24. Tests for circulating neutralising antibodies against interferon-beta will be performed during the study.

ELIGIBILITY:
Inclusion Criteria:

A patient may be included if he/she;

* Is aged between 18 and 55 years (both included).
* Has multiple sclerosis according to the McDonald criteria (McDonald 2001)
* Has a stable disease during the last month period prior to inclusion, and a disability equivalent to EDSS of 5.5 or less (Kurtzke 1983).
* Has shown disease activity defined as at least one relapse or at least one new MRI lesion (T1 enhancing or T2 lesion - ref. McDonald criteria) during the year prior to inclusion.
* Is prepared to and considered able to follow the protocol and to attend the planned visits during the whole study period.
* Is using adequate contraceptive methods and has negative pregnancy test results (female of childbearing potential must).
* Has given written informed consent.

Exclusion Criteria:

A patient has to be excluded if he/she;

* Has received continuous for more than one-week treatment with unsaturated fatty acids (omega-3) within 3 months prior to inclusion in the study.
* Has an active RRMS disease that would strongly be recommended for standard immunomodulatory treatment by the treating neurologist.
* Has received treatment with interferon-beta or glatiramer acetate within 6 months prior to inclusion in the study.
* Has received treatment with lymphoid irradiation, mitoxantrone, cyclophosphamide or long-term glucocorticoids.
* Has received treatment with azathioprine, cyclosporine or other immunosuppressive agents within the year prior to inclusion in the study.
* Has received treatment with glucocorticoids or ACTH within two month prior to inclusion in the study.
* Has experienced a relapse within one month prior to the inclusion in the study.
* Has converted to secondary progressive MS.
* Has suffered from major depression or any other psychiatric disorder that would preclude safe participation in the protocol.
* Has diabetes mellitus.
* Has alcohol or drug abuse.
* Has cardiac insufficiency, cardiomyopathy, significant cardiac dysrhythmia, unstable or advanced ischemic heart disease (NYHA III or IV), or malignant hypertension.
* Has renal insufficiency.
* Has ASAT or ALAT > 2,5 x normal upper limit.
* Has leukopenia < 2500 leukocytes per µl or thrombocytopenia <100 000 thrombocytes per µl.
* Has any systemic disease, which can influence his/her safety and compliance, or the evaluation of the disability.
* Has thromboembolic disease that needs anticoagulative treatment.
* Have formerly shown severe reactions against study drug, interferon-beta or gadolinium (MRI contrast).
* Is breastfeeding or is pregnant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100
Dates: Start 2004-12; Study Completion 2008-07

PRIMARY OUTCOMES:
MRI disease activity measured by the number of new T1-enhancing lesions during the six months of treatment.
MRI disease activity measured by the number of new T1-hypo-intensive lesions (black holes) after 24 months of treatment.

SECONDARY OUTCOMES:
MRI disease activity measured by the number of new T1-enhancing lesions during the first 9 months and the whole study period of 24 months.
Brain atrophy measured by total MRI brain volume at month 6 and month 24
The number of relapses during the first six months and the whole study period of 24 months.
The increase in disability as measured by Expanded Disability Status Scale (EDSS) during the first six months and the whole study period of 24 months.
Changes in the Multiple Sclerosis Functional Composite (MSFC) score during the first six months and the whole study period of 24 months.
MRI disease activity as measured by the number of new or enlarging T2 lesions and enhancing T1 lesions during the first six months and the whole study period of 24 months.
Changes in serum concentrations of mono-unsaturated fatty acids, saturated fatty acids, omega-3- and omega-6 fatty acids during the study.
Changes in immune responses during the first six months and the whole study period of 24 months.
The occurrence of adverse events during the first six months and the whole study period of 24 months.
The occurrence of adverse events during the first three months of interferon-beta 1a (Rebif®) treatment.
The occurrence of neutralising antibodies against interferon-beta 1a (Rebif®) during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Kjell-Morten Myhr, MD, PhD, Study Chair — Dep. of Neurology, Haukeland University Hospital; Antonie G. Beiske, MD, Principal Investigator — Dep. of Neurology, Akershus University Hospital; Harald Hovdal, MD, Principal Investigator — Dep. of Neurology, Trondheim University Hospital; Rune Midgard, MD, PhD, Principal Investigator — Dep. of Neurology, Molde Hospital; Ingrid K. Bjørnå, MD, Principal Investigator — Dep. of Neurology, Buskerud Hospital; Olaf A. Henriksen, MD, Principal Investigator — Dep. of Neurology Nordland Hospital; Jan Schepel, MD, Principal Investigator — Dep. of Neurology Haugesund Hospital; Randi Eikeland, MD, Principal Investigator — Dep. of Neurology Arendal Hospital; Terje Kristensen, MD, Principal Investigator — Dep. of Neurology Fredrikstad Hospital; Halfdan Kierulf, MD, Principal Investigator — Dep. of Neurology Rikshospitalet University Hospital; Frøydis Dalane, MD, Principal Investigator — Dep. of Neurology, Telemark Hospital; Alla Bru, MD, Principal Investigator — Dep. of Neurology, Stavanger University Hospital; Grethe Kleveland, MD, Principal Investigator — Dep. of Neurology, Lillehammer Hospital
Locations (1):
- Department of Neurology, Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Background] Nordvik I, Myhr KM, Nyland H, Bjerve KS. Effect of dietary advice and n-3 supplementation in newly diagnosed MS patients. Acta Neurol Scand. 2000 Sep;102(3):143-9. doi: 10.1034/j.1600-0404.2000.102003143.x. PMID 10987373
- [Derived] Lie IA, Kerklingh E, Wesnes K, van Nederpelt DR, Brouwer I, Torkildsen O, Myhr KM, Barkhof F, Bo L, Vrenken H. The effect of gadolinium-based contrast-agents on automated brain atrophy measurements by FreeSurfer in patients with multiple sclerosis. Eur Radiol. 2022 May;32(5):3576-3587. doi: 10.1007/s00330-021-08405-8. Epub 2022 Jan 3. PMID 34978580
- [Derived] Varhaug KN, Barro C, Bjornevik K, Myhr KM, Torkildsen O, Wergeland S, Bindoff LA, Kuhle J, Vedeler C. Neurofilament light chain predicts disease activity in relapsing-remitting MS. Neurol Neuroimmunol Neuroinflamm. 2017 Nov 28;5(1):e422. doi: 10.1212/NXI.0000000000000422. eCollection 2018 Jan. PMID 29209636
- [Derived] Torkildsen O, Wergeland S, Bakke S, Beiske AG, Bjerve KS, Hovdal H, Midgard R, Lilleas F, Pedersen T, Bjornara B, Dalene F, Kleveland G, Schepel J, Olsen IC, Myhr KM. omega-3 fatty acid treatment in multiple sclerosis (OFAMS Study): a randomized, double-blind, placebo-controlled trial. Arch Neurol. 2012 Aug;69(8):1044-51. doi: 10.1001/archneurol.2012.283. PMID 22507886